CLINICAL TRIAL: NCT07034716
Title: Effects Of Pulsatile and Non-Pulsatile Cardiopulmonary Bypass Flow On Predictors Of Outcome After Coronary Artery Bypass Graft Surgery
Brief Title: Predictors Of Outcome After Coronary Artery Bypass Graft Surgery Using Cardiopulmonary Bypass
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Islam Elbardan, Lecture of anesthesia and surgical intensive care, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0108887
Record Dates: First submitted 2025-06-08; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Clinical Outcomes; Cardiac Surgery; Cardio-pulmonary Bypass
Keywords: Lactate; Perfusion; Central venous saturation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (P): Pulsatile flow will be used during CPB (Experimental): Pulsatile flow will be used during CPB
  Interventions: Procedure: cardiac surgical patients who will undergo isolated elective cardiopulmonary bypass
- Group NP: non-pulsatile perfusion. (Active Comparator): non-pulsatile perfusion during CARDIOPULMONARY BYPASS
  Interventions: Procedure: CORONARY BYPASS SURGERY USING CARDIOPULMONARY BYPASS

INTERVENTIONS:
Procedure: CORONARY BYPASS SURGERY USING CARDIOPULMONARY BYPASS — The study will be conducted on cardiac surgical patients who will undergo isolated elective CABG with nonpulsatile flow during cardiopulmonary bypass
  Arms: Group NP: non-pulsatile perfusion.
Procedure: cardiac surgical patients who will undergo isolated elective cardiopulmonary bypass — The study will be conducted on cardiac surgical patients who will undergo isolated elective CABG with pulsatile flow during cardiopulmonary bypass
  Arms: Group (P): Pulsatile flow will be used during CPB

SUMMARY:
In cardiac operations, high values of blood lactate have been associated with bad outcomes if detected both during CPB and at the arrival in the intensive care unit (ICU) in adult patients. Many studies highlighted the potential role of hyperlactatemia on admission to the ICU as a marker for adverse outcome, and one study linked hyperlactatemia during CPB with postoperative morbidity and mortality. Evidence that both CENTRAL VENOUS SATURATION (ScVO2) and blood lactates during CPB are potential early predictors of morbidity and mortality in adult cardiac operations are still lacking.

ELIGIBILITY:
Inclusion Criteria:

cardiac surgical patients who will undergo isolated elective CABG and fulfill these criteria:

1. Aged 18 years or above.
2. Operated with cardiopulmonary bypass.

Exclusion Criteria:

1. Preoperative lactate level greater than 3 mmol/l.
2. Redo surgery.
3. If the patient will be reoperated during the study time.
4. Preoperative hemoglobin level less than 10 mg/dl.
5. Ejection fraction (EF) of <30%.
6. Renal impairment.
7. Liver impairment.
8. History of stroke and significant carotid artery stenosis.
9. Chronic obstructive or restrictive lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
effects of pulsatile versus non-pulsatile perfusion methods in CABG surgeries on arterial lactate level. | 24 hour
  Arterila Lactate values (mmol/L).
effects of pulsatile versus non-pulsatile perfusion methods in CABG surgeries on saturation of central venous blood. | 24 hour
  saturation of central venous blood (percentage)

SECONDARY OUTCOMES:
The duration of mechanical ventilation (hours). | 24 hour
Length of ICU stay (days) | 24 hour
Occurrence of major morbidity | 72 hours
  The occurrence of at least one in-hospital morbidity with or without in-hospital mortality. (Stroke, seizures, myocardial ischemia, low cardiac output state, post-perfusion syndrome, acute kidney injury, pancreatitis, acute hepatitis, and any other complication will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: LECTURER OF ANESTHESIA AND SURGICAL INTENSIVE CARE, Principal Investigator — University of Alexandria